CLINICAL TRIAL: NCT01114295
Title: Comparative Effectiveness of Wireless Capsule Endoscopy and Dual Energy, Phase CT Enterography in the Evaluation of Overt Obscure GI Bleeding
Brief Title: Computed Tomography Enterography (CTE) Versus Capsule Endoscopy for Overt, Obscure Gastrointestinal (GI) Bleeding
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped before the first patient was enetered due to logistical issues and lack of funding.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, John Robinson Saltzman, MD, Director of Endoscopy, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTE vs Capsule 2010
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Recurrent Gastrointestinal Bleeding
Keywords: overt; obscure; gastrointestinal; bleeding; hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overt Obscure Gastrointestinal Bleeders (Experimental): The only cohort in this study are those patients identified as having overt, obscure gastrointestinal bleeding who will then undergo CE or CTE.
  Interventions: Device: Capsule Endoscopy; Radiation: CT Enterography

INTERVENTIONS:
Device: Capsule Endoscopy — Prior to the test, patients will be on a clear liquid diet for 24 hours and will have undergone an overnight fast. If a clear liquid diet is not possible, some patients may undergo a bowel preparation the day before the procedure. On the morning of the test, patients will swallow a video capsule with water. Clear liquids will be permitted after 2 hours, and a light meal permitted 4 hours after swallowing the capsule, if appropriate. No medications will be allowed 2 hours before the procedure and drugs that can delay gastric emptying will be avoided until the study is complete. At 8 hours after ingestion, the sensor array and recorder/battery belt pack will be disconnected and the data will be downloaded onto a computer equipped with software for image viewing. Images are sent through 8 skin electrodes to the recorder, stored and viewed on a RAPID workstation. At the end of the recording, the video is transferred to a computer for analysis.
Radiation: CT Enterography — CT enterography at the Brigham and Women's hospital is performed by using intravenous iodinated contrast material (Ultravist 300) and a neutral oral-enteric contrast material containing methylcellulose (Volumen). During scanning, 150 mL of nonionic intravenous contrast medium will be administered at a rate of 3mL/sec and the imaging conducted 40 and 70 seconds after the administration of the intravenous contrast medium. All imaging will be performed on a Dual-Energy multi-detector row CT scanner, Somatom Definition (Siemens Healthcare, Forcheim, Germany). Two independent X-ray tube/detector system will be used for image acquisition. One tube operates at 140 kV and the other at 80 kV . Slice collimation will be 0.6 mm and images reconstructed at 3 mm thickness with 3 mm reconstruction intervals. Coronal and sagittal images will be reconstructed at 3 mm thickness with 3 mm increments. Images will be reviewed by a radiologist experienced in the interpretation of CT enterography.

SUMMARY:
Up to 5% of patients with recurrent gastrointestinal (GI) bleeding remain undiagnosed by upper endoscopy and colonoscopy, the presumed source of bleeding in these patients being the small intestine. These patients fall under the category of "obscure gastrointestinal bleeding," and frequently require an extensive diagnostic work-up.

Obscure gastrointestinal bleeding (OGIB) refers to bleeding undiagnosed by upper endoscopy and colonoscopy. In 40-70% of cases of OGIB, a bleeding lesion is localizable to the small bowel. In OGIB, capsule endoscopy (CE) has a diagnostic yield of 40-80%, and has demonstrated diagnostic superiority to push enteroscopy, barium studies, angiography, CT angiography, and routine abdominal CT scan. When CE is non-diagnostic, however, the subsequent diagnostic algorithm is not well-defined. There is currently no established role for cross-sectional imaging for this indication. CT enterography (CTE) combines the spatial and temporal resolution of CT with an orally administered neutral enteric contrast material that permits detailed visualization of the small bowel. Unlike other imaging modalities such as nuclear medicine techniques and catheter angiography, CT is less labor-intensive, more readily available, and provides precise anatomic localization. A novel OGIB-protocol available at Brigham and Women's Hospital for CTE utilizes a dual-phase, dual energy technique that obtains images at two time points to better identify active bleeding in the mesentery. We, the investigators, plan to prospectively study an algorithm that employs CTE and compare to capsule endoscopy to investigate the effectiveness of both modalities and to evaluate the potential role of CTE in OGIB.

The goal of our study is to determine observationally the contribution of both CE and the new protocol for CTE to the evaluation and management of overt obscure GI bleeding and accordingly revise the clinical algorithm.

We hypothesize that CTE will be as or more effective than CE at identifying culprit lesions in overt, obscure gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with signs and symptoms of "overt, obscure GI bleeding" including hematemesis, melena, and hematochezia within the past 14 days with negative endoscopic evaluation (including upper endoscopy for hematemesis, and both upper and lower endoscopy for hematochezia) despite clinical evidence of GI bleeding.

Exclusion Criteria:

* Known renal insufficiency (or blood Creat >1.5 or estimated glomerular filtration rate [eGFR]<60)
* Allergy to iodinated intravenous (IV) contrast media
* Swallowing difficulties
* Known small bowel strictures
* Suspected bowel obstruction
* Under the age of 18
* Unable to give consent
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Detection of an actively bleeding lesion or lesion believed to be causing bleeding symptoms. | 2-3 days
  Patients enrolled in the study will undergo either capsule endoscopy or CT enterography first, and this decision will generally be based on which test the clinical providers have already scheduled or availability of testing as is done with routine clinical care. The results of each the test will be read by an experienced gastroenterologist or radiologist respectively. These reviewers will be blinded to the results of any other diagnostic studies. The patient will then undergo the second test.

SECONDARY OUTCOMES:
Contribution of diagnostic test to clinical management | 30 days
  We will assess whether either CT or CTE changes managemet based on findings
Overall cost of evaluation | 30 days
  We will assess the cost of each test and cost based on findings
Adverse events | 30 days
  We will measure any and all adverse outcomes based on CT or CTE for the month following whichever study is performed last.

CONTACTS AND LOCATIONS:
Overall Officials: John Saltzman, MD, Principal Investigator — Brigham and Women's Hospital